CLINICAL TRIAL: NCT06414798
Title: A First-in-Human Single Ascending Dose, Mass Balance, and Food Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ABBV-1088 in Healthy Adult Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of ABBV-1088 Oral Dose in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: M24-929
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; ABBV-1088

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Group 1- ABBV-1088 Dose A (Experimental): Participants will receive single dose of ABBV-1088 dose A on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 1- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088
- Group 2- ABBV-1088 Dose B (Experimental): Participants will receive single dose of ABBV-1088 dose B on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 2- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088
- Group 3- ABBV-1088 Dose C (Experimental): Participants will receive single dose of ABBV-1088 dose C on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 3- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088
- Group 4- ABBV-1088 Dose D (Experimental): Participants will receive single dose of ABBV-1088 dose D on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 4- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088
- Group 5- ABBV-1088 Dose E (Experimental): Participants will receive single dose of ABBV-1088 dose E on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 5- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088
- Group 6- ABBV-1088 Dose F (Experimental): Participants will receive single dose of ABBV-1088 dose F on day 1
  Interventions: Drug: Drug: ABBV-1088
- Group 6- Placebo (Experimental): Participants will receive single dose of placebo day 1
  Interventions: Drug: Drug: Placebo for ABBV-1088

INTERVENTIONS:
Drug: Drug: ABBV-1088 — • Oral Capsule
  Arms: Group 1- ABBV-1088 Dose A; Group 2- ABBV-1088 Dose B; Group 3- ABBV-1088 Dose C; Group 4- ABBV-1088 Dose D; Group 5- ABBV-1088 Dose E; Group 6- ABBV-1088 Dose F
Drug: Drug: Placebo for ABBV-1088 — • Oral Capsule
  Arms: Group 1- Placebo; Group 2- Placebo; Group 3- Placebo; Group 4- Placebo; Group 5- Placebo; Group 6- Placebo

SUMMARY:
This study will assess the single dose safety, tolerability and pharmacokinetic properties of ABBV-1088 in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG

Exclusion Criteria:

* History of cardiac disease, including congenital structural/conduction abnormalities, cardiomyopathy, myocardial infarction, cardiac arrhythmia.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, chronic GERD, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection, etc.].
* History of suicidal ideation within one year prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at Screening, or any history of suicide attempts within the last two years.
* History of any clinically significant neurological, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-1088 | Up to approximately 11 days
  Cmax of ABBV-1088
Time to Cmax (Tmax) of ABBV-1088 | Up to approximately 11 days
  Tmax of ABBV-1088
Terminal Phase Elimination Rate Constant (Beta) of ABBV-1088 | Up to approximately 11 days
  Terminal phase elimination rate constant (beta) of ABBV-1088
Terminal Phase Elimination Half-Life (t1/2) of ABBV-1088 | Up to approximately 11 days
  Terminal phase elimination half-life of ABBV-1088
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-1088 | Up to approximately 11 days
  AUCt of ABBV-1088
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-1088 | Up to approximately 11 days
  AUCinf of ABBV-1088
Number of Participants With Adverse Events (AEs) | Up to Day 32
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 264249, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-929